CLINICAL TRIAL: NCT02014779
Title: Internet-Based Relapse Prevention With Therapist Support vs Face to Face Therapy at an Employee Assistance Program: A Randomized Controlled Non-inferiority Trial
Brief Title: Internet-Based Relapse Prevention vs Face to Face Therapy at an Employee Assistance Program
Acronym: FoBeMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 1 participant recruited to study. Qs addressed in other ongoing studies.
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1391-31/5
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Alcohol Abuse; Alcohol Addiction
Keywords: Randomized Controlled Trial; Alcohol; Internet; Internet based therapy; Cognitive behavioral therapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eChange web-based relapse prevention (Experimental): A relapse intervention program consisting of 14 modules. Patients will have access to therapist support through an internal secure messaging system.
  Interventions: Behavioral: eChange
- Face-to-face therapy (Active Comparator): Face-to-face psychotherapy, consisting of 20 sessions. The content will be vary for different therapists, but all have an evidence-based approach to therapy
  Interventions: Behavioral: Face-to-face therapy

INTERVENTIONS:
Behavioral: eChange — A web-based relapse intervention program consisting of 14 modules. The patient will have access to therapist support through a secure messaging system
  Arms: eChange web-based relapse prevention
Behavioral: Face-to-face therapy — Face-to-face psychotherapy, consisting of 20 sessions. The content will be different for different therapists, but all have an evidence based approach to therapy
  Arms: Face-to-face therapy

SUMMARY:
Objectives: This study will evaluate the efficacy of internet-based relapse prevention with therapist support, as compared to face-to-face therapy at an employee assistance program. The design is a two-armed randomized controlled design, and outcomes are measured in terms of changes in problematic alcohol use, as well as depression and quality of life.

Method: Participants with problematic alcohol use who, after an initial evaluation consisting of five face-to-face sessions with a licensed psychologist where alcohol and collateral problems are extensively assessed, are recommended treatment for problematic alcohol use. Consenting participants will be randomized into one of two groups: 1. Internet delivered relapse prevention with therapist support or 2. Face-to-face therapy. Outcomes on alcohol use, depression and quality of life as well as information on user satisfaction will be gathered post treatment. Follow up will be at 3, 6 and 12 months after completion.

Our hypothesis is that the internet-based program with therapist support and the face-to-face therapy will be equally effective in reducing alcohol use (non-inferiority).

ELIGIBILITY:
Inclusion Criteria:

Problematic alcohol use and having been recommended psychotherapy by the assessing psychologist.

Exclusion Criteria:

Inadequate Swedish language skills No Internet access Reading and/or writing difficulties Major depression Current suicidal thoughts and/or plans Primary problematic drug use PTSD-related problems Psychosis Cognitive disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Identification Test (AUDIT) | Post, 3, 6 and 12 months
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems)

SECONDARY OUTCOMES:
Time Line Follow Back (TLFB) | Post, 3, 6 and 12 months
  Change in total TLFB score, as a summarized measure of alcohol consumption
Montgomery Asberg Depression Rating Scale - Self report (MADRS-S) | Post, 3, 6 and 12 months
  Change in total MADRS-S score, as a summarized measure of depression
World Health Quality of Life Scale (WHOQOL-BREF) | Post, 3, 6 and 12 months
  Change in total WHOQOL-BREF score, as a summarized measure of quality of life

OTHER OUTCOMES:
Drug Use Identification Test (DUDIT) | Post, 3, 6 and 12 months
  Change in total DUDIT score, as a summarized measure of drug (including alcohol consumption and alcohol-related problems)
Biological tests for alcohol markers | Post
  Biological marker outcomes post-treatment. B-PEth and CDT.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Stockholm, Sweden